CLINICAL TRIAL: NCT05959278
Title: Pilot Feasibility of App-supported Vestibular Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Ben-Gurion University of the Negev (Other); Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Yoav Gimon, Head of the dizziness clinic, Sheba Hospital, University of Haifa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: SHEBA-23--957622-AW-CTIL
Record Dates: First submitted 2023-07-06; First posted 2023-07-25 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Vestibular Disorder
MeSH Terms: conditions — Vestibular Diseases | interventions — Amyloid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Vestibular rehabilitation - initially supported by the app (Experimental): First two and a half weeks - conventional vestibular rehabilitation supported by an app Second two and a half weeks - conventional vestibular rehabilitation without an app
  Interventions: Other: App for vestibular rehabilitation
- Group 2 - Vestibular rehabilitation - initially without the support of the app (Experimental): First two and a half weeks - conventional vestibular rehabilitation without an app Second two and a half weeks - conventional vestibular rehabilitation supported by an app
  Interventions: Other: App for vestibular rehabilitation

INTERVENTIONS:
Other: App for vestibular rehabilitation — This app is a platform for performing conventional vestibular rehabilitation remotely

SUMMARY:
The primary goal of the study is to examine the feasibility of accompanying vestibular practice supported by a phone app for vestibular rehabilitation. Feasibility will be established using the following parameters: (1) the User Satisfaction Evaluation Questionnaire (USEQ) (2) a custom-made questionnaire to collect feedback from participants, and (3) compliance measurements derived from app usage. The secondary goal of the study is to examine the effect of practice supported by the app on balance and anxiety indices. These will be measured using the following parameters: (1) Instrumented Timed Up and Go Test (iTUG), (2) Dizziness Handicap Inventory (DHI), (3) State-Trait Anxiety Inventory (STAI). The third goal is to assess the correlation between balance function (iTUG) and anxiety (STAI).

A randomized crossover pilot study will be conducted with 24 participants. During the study, each group will undergo two and a half weeks of conventional vestibular rehabilitation and two and a half weeks of app-supported vestibular rehabilitation. Measurement sessions will be conducted at three-time points: upon enrollment in the study (T0), after two and a half weeks (T1), and at the end of the study (T2).

ELIGIBILITY:
Inclusion Criteria:

Participants that will meet the following inclusion criteria were recruited to the study:

1. between the ages of 18-75;
2. diagnosis of vestibular dysfunction;
3. fluent in Hebrew;
4. own an Android smart-phone

Exclusion Criteria:

Exclusion criteria for the study group will be as follows:

1. a medical condition that prevents participant from performing home vestibular rehabilitation practice - such as orthopedic, neurological, cardiac, visual impairment;
2. individuals with dizziness who already have been given a home vestibular rehabilitation exercise program;
3. diagnosis of central vestibular disorder due to brain structural damage.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-07-16 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Instrumented Timed Up and Go Test (iTUG) (Change) | In each of the measurement sessions - baseline, after two and a half weeks, and after five weeks
  The Timed Up and Go Test (TUG) examine functional balance
  The investigators will use the Instrumented Timed Up and Go Test (iTUG), for a combination of qualitative and quantitative assessment for this test. For the measurement, the investigators will use Opal (APDM) sensors.
  Measurements will be repeated three times to determine whether any changes have occurred during the rehabilitation process.
State-Trait Anxiety Inventory (STAI) (Change) | In each of the measurement sessions - baseline, after two and a half weeks, and after five weeks
  The STAI is a self-reported questionnaire designed to examine a person's general and current anxiety levels. The investigators will use this questionnaire to better distinguish between the participant's general and momentary anxiety to assess vestibular rehabilitation's effect on anxiety levels.
  This is a questionnaire with a numerical score between 40-160, a higher score indicates more anxiety.
  Measurements will be repeated three times to determine whether any changes have occurred during the rehabilitation process.
Dizziness Handicap Inventory (DHI) (Change) | In each of the measurement sessions - baseline, after two and a half weeks, and after five weeks
  The DHI is a 25-items questionnaire designed to assess the impact of dizziness on everyday life in people with vestibular disorders.
  This is a questionnaire with a numerical score between 0-100; a higher score indicates a higher level of handicap.
  Measurements will be repeated three times to determine whether any changes have occurred during the rehabilitation process.
Custom-made questionnaire | After two and a half weeks of using the application
  The questionnaire includes questions regarding the user's experience with the application.
  The investigators will use the questionnaire to get the participants' feedback on using the app and to examine the feasibility of using the app in vestibular rehabilitation.
  This questionnaire mostly includes open-ended questions in free text and a part that includes questions with a numerical rating between 5-30. A higher score indicates a better user experience in the app.
User Satisfaction Evaluation Questionnaire (USEQ) | After two and a half weeks of using the application
  The investigators will use the questionnaire to get the participants' feedback on the use of the app, and to examine the feasibility of using the app in vestibular rehabilitation
  This is a questionnaire with a numerical score between 5-30; a higher score indicates a higher satisfaction level.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Wolfovitz, Dr., Principal Investigator — Sheba Meical Center
Locations (1):
- Sheba Hospital, Ramat Gan, Center, Israel

REFERENCES:
- [Background] Hall CD, Herdman SJ, Whitney SL, Anson ER, Carender WJ, Hoppes CW, Cass SP, Christy JB, Cohen HS, Fife TD, Furman JM, Shepard NT, Clendaniel RA, Dishman JD, Goebel JA, Meldrum D, Ryan C, Wallace RL, Woodward NJ. Vestibular Rehabilitation for Peripheral Vestibular Hypofunction: An Updated Clinical Practice Guideline From the Academy of Neurologic Physical Therapy of the American Physical Therapy Association. J Neurol Phys Ther. 2022 Apr 1;46(2):118-177. doi: 10.1097/NPT.0000000000000382. PMID 34864777
- [Background] Kim KJ, Gimmon Y, Millar J, Brewer K, Serrador J, Schubert MC. The Instrumented Timed "Up & Go" Test Distinguishes Turning Characteristics in Vestibular Hypofunction. Phys Ther. 2021 Jul 1;101(7):pzab103. doi: 10.1093/ptj/pzab103. PMID 33774661
- [Background] Meldrum D, Burrows L, Cakrt O, Kerkeni H, Lopez C, Tjernstrom F, Vereeck L, Zur O, Jahn K. Vestibular rehabilitation in Europe: a survey of clinical and research practice. J Neurol. 2020 Dec;267(Suppl 1):24-35. doi: 10.1007/s00415-020-10228-4. Epub 2020 Oct 13. PMID 33048219
- [Background] Polensek SH, Tusa RJ, Sterk CE. The challenges of managing vestibular disorders: a qualitative study of clinicians' experiences associated with low referral rates for vestibular rehabilitation. Int J Clin Pract. 2009 Nov;63(11):1604-12. doi: 10.1111/j.1742-1241.2009.02104.x. PMID 19832817
- [Background] Rosiak O, Krajewski K, Woszczak M, Jozefowicz-Korczynska M. Evaluation of the effectiveness of a Virtual Reality-based exercise program for Unilateral Peripheral Vestibular Deficit. J Vestib Res. 2018;28(5-6):409-415. doi: 10.3233/VES-180647. PMID 30714985
- [Background] Whitney SL, Alghwiri AA, Alghadir A. An overview of vestibular rehabilitation. Handb Clin Neurol. 2016;137:187-205. doi: 10.1016/B978-0-444-63437-5.00013-3. PMID 27638071